CLINICAL TRIAL: NCT04508920
Title: A Survey to Assess Effects of the Covid-19 Pandemic on Symptomatology, Treatment and Medical Care for Cardiovascular Patients
Brief Title: A Survey to Assess Effects of Covid-19 on Cardiovascular Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro en Insuficiencia Cardiaca, Mexico (Other)
Collaborators: Instituto Nacional de Cardiologia Ignacio Chavez (Other); Medica Sur Clinic & Foundation (Other)
Responsible Party: Principal Investigator, EDUARDO CHUQUIURE-VALENZUELA MD MSc FACC, Principal investigator, Centro en Insuficiencia Cardiaca, Mexico
Other Study IDs: 20-1156
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Diseases; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Basal: All adults (age >18 years), both gender, Heart failure patients (european society of cardiology ) criteria, sign consent.
  A survey to access information about symptomatology, treatment, and medical care in period may 15 to june 15, 2019 ( without covid-19 )
  Interventions: Other: Symptomatology, Treatment. daily Activities and Anxiety for Cardiovascular patients Survey (STRATA)
- Ourbreak: All adults (age >18 years), both gender, Heart failure patients (european society of cardiology ) criteria, sign consent.
  A survey to access information about symptomatology, treatment, and medical care in period may 15 to june 15, 2020 ( ongoing covid-19 )
  Interventions: Other: Symptomatology, Treatment. daily Activities and Anxiety for Cardiovascular patients Survey (STRATA)

INTERVENTIONS:
Other: Symptomatology, Treatment. daily Activities and Anxiety for Cardiovascular patients Survey (STRATA) — Interventions were recorded in two groups of patients, who were randomly selected, in two different periods of time. The basal group was intervened from 15 May to 15 June 2019, a pandemic-free period. The outbreak group from 15 May to 15 June 2020, corresponding to increased activity of contagiousness and mortality associated with COVID-19, in general population in Mexico14 Basal measurement was performed in a face to face method. In Outbreak period, under social isolation conditions, patients were evaluated by telephone. The assessments were performed out by medical staff with specialized training, with evaluations to which patients were accustomed by regular cohort assessments. The questions were ordered and systematized in a patient evaluation, care, and follow-up guide (appendix). A causality association question of emotional distress perception was added. We recorded mortality and rehospitalization
  Other Names: STRATA survey

SUMMARY:
The design included 152 patients with confirmed heart failure (HF) evaluated in two different periods of time: a baseline before the outbreak, and other during the outbreak of which 76 patients were randomized in each group. A care and follow-up guide was used as an instrument through a face-to-face survey (baseline group) and telemedicine (group outbreak). The primary outcome was the comparison of functional class modification observed in patients

DETAILED DESCRIPTION:
Population and Data Sources All patients included, confirmed diagnosis of HF, according with the ESC guidelines criteria, both genders, above 18 years, who agreed to participate. All HF outpatients belonged to an open follow-up cohort of the HF clinic of the National Institute of Cardiology of Mexico, which started enrollment since September 2016. Periodic determinations were planned, clinical, functional, therapeutic evaluations, and emotional distress. The present design is a nested comparative analysis through a care and follow-up guide to HF patients.

Data collection and outcomes Interventions were recorded in two groups of patients, who were randomly selected, in two different periods of time. The basal group was intervened from 15 May to 15 June 2019, a pandemic-free period. The outbreak group from 15 May to 15 June 2020, corresponding to increased activity of contagiousness and mortality associated with COVID-19, in general population in Mexico.

Basal measurement was performed in a face to face method. In Outbreak period, under social isolation conditions, patients were evaluated by telephone. The assessments were performed out by medical staff with specialized training, with evaluations to which patients were accustomed by regular cohort assessments. The questions were ordered and systematized in a patient evaluation, care, and follow-up guide . A causality association question of emotional distress perception was added. Investigators recorded mortality and rehospitalization.

The primary outcome was comparison of functional class modification, secondary outcomes were Clinical alterations related to HF worsening, Therapeutic modifications, Daily physical activities, and Self-perception of health status.

The protocol conducted to hypothesize that the clinical alarm data reported by patients, in an alternative in-home model, with tele-medical assistance, is a useful tool in follow-up, as in detecting therapeutic performances, and associated with the HF deterioration.

Protocol was approved by the ethics and investigational committees. All patients previously signed informed consent. Additionally, prior to the telephone survey, a verbal assent was requested. Absolute confidentiality of all patient data was declared.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of HF, according with the ESC guidelines criteria
* both genders,
* above 18 years,
* agreed to participate

Exclusion Criteria:

* Impediment to contacting patients
* marked physical impairment
* cognitive impairment that prevents optimal interrogation
* Cultural barriers involving communication limitation (languages, dialects, reading and writing)
* Patient doesn't want to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HF outpatients belonged to an open follow-up cohort of the HF clinic of the National Institute of Cardiology of Mexico, which started enrollment since September 2016.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
NYHA class deterioration | 1 year
  NYHA class modification in the last four weeks. Basal and follow-up measures: Basal on June 2020. Follow up: every three months and a year (June 2021). NYHA Scale: Minimum: 1 to maximum :4

SECONDARY OUTCOMES:
Dyspnea deterioration | 1 year
  physiological parameter to worsening of shortness of breath perception, in last four weeks. Basal and follow-up measures: Basal on June 2020. Follow up: every three months and a year (June 2021).Dichotomic scale presence or absence
Paroxysmal nocturnal dyspnea deterioration | 1 year
  Physiological parameter to worsening of dyspnea that suddenly occurs to decubitus, in last four weeks. Basal and follow-up measures: Basal on June 2020. Follow up: every three months and a year (June 2021). Dichotomic scale presence or absence.
Edema | 1 year
  Physiological parameter to worsening of quantification of swollen ankles in both pelvic limbs, in last four weeks. Basal and follow-up measures: Basal on June 2020. Follow up: every three months and a year (June 2021). Dichotomic scale presence or absence
Daily activities In the last four weeks? Please, mention if you a perceived limitation on : Walking deterioration | 1 year
  a perceived limitation on walking more 500 meters, in last four weeks. Basal and follow-up measures: Basal on June 2020. Follow up: every three months and a year (June 2021). Dichotomic scale presence or absence.

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO CHUQUIURE-VALENZUELA, MD, Principal Investigator — Centro en insuficiencia cardiaca
Locations (1):
- Centro de Insuficiencia Cardiaca Instituto Nacional de Cardiologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
IPD PLAN Eduardo Chuquiure-Valenzuela is Principal investigator, conceptual protocol designer, performed statistics, write manuscript and draft corrections.
  Alan Fuentes-Mendoza, Emmanuel Tapia-López, Daniel García-Romero Elyz Cortez-Lopez and Alejandra Marin-Sanchez, collaborate in clinical, research and analysis activities for CENTRO EN INSUFICIENCIA CARDIACA, Also, they assist in telephone interviews, writing of the manuscript. performed and checked statistics, co- writer, and draft corrections.
  Laura Rodríguez Chávez, Nilda Espíndola Zavaleta, Gerardo Vieyra Herrera, and Enrique Lopez Mora, are affiliated cardiologists, who participate in the draft revision for publication.
Supporting Information: Study Protocol, ICF
Time Frame: august 1, 2021 to december 30,2021
Access Criteria: open access
URL: http://cardiologia.org.mx

REFERENCES:
- [Background] Cowie MR, Mosterd A, Wood DA, Deckers JW, Poole-Wilson PA, Sutton GC, Grobbee DE. The epidemiology of heart failure. Eur Heart J. 1997 Feb;18(2):208-25. doi: 10.1093/oxfordjournals.eurheartj.a015223. No abstract available. PMID 9043837
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Judd SE, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Mackey RH, Magid DJ, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER 3rd, Moy CS, Mussolino ME, Neumar RW, Nichol G, Pandey DK, Paynter NP, Reeves MJ, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014 Jan 21;129(3):e28-e292. doi: 10.1161/01.cir.0000441139.02102.80. Epub 2013 Dec 18. No abstract available. PMID 24352519
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Hawkins NM, Jhund PS, McMurray JJ, Capewell S. Heart failure and socioeconomic status: accumulating evidence of inequality. Eur J Heart Fail. 2012 Feb;14(2):138-46. doi: 10.1093/eurjhf/hfr168. PMID 22253454
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Inciardi RM, Lupi L, Zaccone G, Italia L, Raffo M, Tomasoni D, Cani DS, Cerini M, Farina D, Gavazzi E, Maroldi R, Adamo M, Ammirati E, Sinagra G, Lombardi CM, Metra M. Cardiac Involvement in a Patient With Coronavirus Disease 2019 (COVID-19). JAMA Cardiol. 2020 Jul 1;5(7):819-824. doi: 10.1001/jamacardio.2020.1096. PMID 32219357
- [Result] Anderson JL, Heidenreich PA, Barnett PG, Creager MA, Fonarow GC, Gibbons RJ, Halperin JL, Hlatky MA, Jacobs AK, Mark DB, Masoudi FA, Peterson ED, Shaw LJ. ACC/AHA statement on cost/value methodology in clinical practice guidelines and performance measures: a report of the American College of Cardiology/American Heart Association Task Force on Performance Measures and Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Jun 3;63(21):2304-22. doi: 10.1016/j.jacc.2014.03.016. Epub 2014 Mar 27. No abstract available. PMID 24681044

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT04508920/Prot_ICF_000.pdf